CLINICAL TRIAL: NCT05047913
Title: Comprehensive Evaluation of Tumor Oxygenation, Metabolism and Blood Supply of High Grade Glioma and Cervical Cancers Using Dynamic FAZA PET and Multiparametric MR
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0285; NCI-2021-10764 (Other: NCI-CTRP Clinical Trials Processing Registry)
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor; Cervical Cancer
MeSH Terms: conditions — Brain Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FTX (Experimental): The radioactive tracer (FAZA)
  Interventions: Drug: 18F-FTX

INTERVENTIONS:
Drug: 18F-FTX — Given By IV

SUMMARY:
Primary Objectives To investigate the relationship between dynamic MRI, brain tumor perfusion (DSC) and permeability (DCE), and dynamic 18F-FAZA PET uptake.

Secondary Objectives To investigate the relationship between tumors with greater hypoxia defined by qBOLD and 18F-FAZA PET and pathological features including proportionate necrosis, Ki-67 and IDH mutation status

To investigate the correlation between the hypoxic tumor region delineated using 18F-FAZA PET and qBOLD

ELIGIBILITY:
Inclusion Criteria:

Glioma Cohort

* Adult (> 18 years old) patients with newly diagnosed or recurrent high grade glioma with newly confirmed pathology (within 1 month)
* Able to provide informed consent
* No contraindications to MRI with gadolinium contrast or 18F-FAZA PET

Cervical Cohort

* Adult (>18 years old) female with newly diagnosed cervical cancer
* Able to provide informed consent
* Receiving surgery, radiotherapy or chemotherapy
* No contraindication to MRI with gadolinium contrast or 18F-FAZA PET

Exclusion Criteria:

Glioma Cohort

* Prior nephrectomy or planned nephrectomy.
* Prior brain radiation within 30 days.
* Pregnant or lactating women: Pregnant women are excluded from this study because the effects of 18F-FAZA in pregnancy are not known. A urine or serum pregnancy test will be performed before enrollment after informed consent is obtained. The pregnancy test is part of SOC before imaging.
* Lactation should be suspended for at least two days following the administration of 18F-FAZA to the mother, because of the unknown but potential risk for adverse events in nursing infants secondary to administration of the radionuclide to a lactating woman.
* Subjects with contraindications to the use of 18F-FAZA including confirmed allergy.
* Patients with a body weight of 400 pounds or more, or a BMI which precludes their entry into the bore of the PET-MRI scanner, because the findings will probably be compromised in image quality with PET-MRI.
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the investigator may significantly interfere with study compliance.

Cervical Cohort

* Prior nephrectomy or planned nephrectomy.
* Pregnant or lactating women: Pregnant women are excluded from this study because the effects of 18F-FAZA in pregnancy are not known. A urine or serum pregnancy test will be performed before enrollment after informed consent is obtained. The pregnancy test is part of SOC before imaging.
* Lactation should be suspended for at least two days following the administration of 18F-FAZA to the mother, because of the unknown but potential risk for adverse events in nursing infants secondary to administration of the radionuclide to a lactating woman.
* Subjects with contraindications to the use of 18F-FAZA including confirmed allergy.
* Patients with a body weight of 400 pounds or more, or a BMI which precludes their entry into the bore of the PET-MRI scanner, because the findings will probably be compromised in image quality with PET-MRI and MRI.
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To correlate the relationship between dynamic MRI (tumor perfusion (DSC) and permeability (DCE)) and dynamic 18F-FAZA PET uptake. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT05047913/ICF_000.pdf